CLINICAL TRIAL: NCT03940157
Title: Faith and Community in Action: Increasing Awareness and Management of Depression in African American Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Urban League of Greater Madison (Unknown); African American Council of Churches Madison (Unknown); Second Baptist Church (Unknown); YWCA of Madison (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0129; A545000 (Other: UW Madison); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison)
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Depression; Awareness; Self-management
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: All participants will be exposed to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oh Happy Day Class - Still I Rise (Experimental): The Oh Happy Day Class-Still I Rise (OHDC-SIR) is a one-time, 4-hour class focused on awareness of depression and healthy self-management strategies ( a workbook is created with the class content). The class is offered in non clinical setting, but will be delivered in a classroom setting at the University. The class will be taught by the PI Dr. Ward, who is an associate professor and licensed psychologist, and Dr. Ward's research program manager, Lucretia Sullivan-Wade.
  Interventions: Behavioral: Oh Happy Day Class - Still I Rise

INTERVENTIONS:
Behavioral: Oh Happy Day Class - Still I Rise — one-time, 4-hour class focused on awareness of depression and healthy self-management strategies

SUMMARY:
Specific Aims/Study Objectives:

1. Evaluate acceptability and implementation of the "Oh Happy Day: Still I Rise Class," which comprise a one-time 4-hour class in which participants will learn about depression with the goal of increasing knowledge of depression and self-management of depression with use of a guided class and self-help workbook. Measures of acceptability will include class attendance, completion of workbook activities and satisfaction. Measures of implementation will include satisfaction, class enrollment, fidelity in delivery of class content, and cost analysis.

2) Evaluate participants' knowledge of depression pre-and immediate post-class, and 3-months post class. Measure: depression quiz. The investigators hypothesize participants will show increased knowledge of depression pre -and post-class.

3) Examine effectiveness of the Oh Happy Day Class- Still I Rise (OHDC-SIR) in prevention of depression and 3- months' post- class. Measure, Patient Health Questionnaire - ( PHQ-9)

4) Examine effectiveness of OHDC-SIR in reducing symptoms of depression 3- months' post- class. Measure, PHQ-9. The investigators hypothesize the OHDC-SIR will result in reduction in depressive symptoms 3- months' post-class.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a major public health concern and is quickly approaching the status of a global public health crisis. According to the World Health Organization, by 2020 MDD will be the leading cause of disability globally. In the US an estimated 9.0% of adults report symptoms for current MDD (i.e., during the preceding 2 weeks). It is well documented that women (4.0%) are significantly more likely to report and be diagnosed with MDD compared to men (2.7%) NIMH, 20017). In addition, health disparities research examining MDD show African Americans evidence higher prevalence of depression (4.0%) compared to Whites (3.1%) and African Americans report more chronic MDD and associated disability than do Whites (56.5% vs. 38.6%; Williams et al., 2007). Despite being burdened by MDD, African Americans evidences low seeking of professional help. However, they highly rely on religious coping. This, it is important to work in partnership with African American clergy and African Americans in community based research to create programs that are more aligned with their cultural and religious beliefs.

Investigators propose using a one-group (OHDC-SIR) non-randomized observational trial and a sample of 100 African American men and women participants (age 25 and older) with measures at baseline, immediately at the end of the class, and 3- months' post-class. The total duration of the study is 4 months.

ELIGIBILITY:
Inclusion Criteria:

* African American male or female
* Age 25 and older
* Residence in the state of Wisconsin
* With or without depression

Exclusion Criteria:

* Self-report of a psychotic disorder such as

  * schizophrenia
  * bipolar disorder
* Cognitive disorder such as dementia
* Presently experiencing suicidal ideations.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PhQ-9) | 4 months
  Patient Health Questionnaire (PHQ-9 is a depression measure. PHQ-9 is a self-administered (5 minutes completion time) depression scale, which scores each of the 9 DSM-IV (Diagnostic and Statistical Manual-IV) criteria as "0" (not at all) to "3" (nearly every day). A PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores are summed, and scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively. In addition to making criteria-based diagnoses of depressive disorders, the PHQ-9 is also a reliable and valid measure of depression severity. These characteristics plus its brevity make the PHQ-9 a useful clinical and research tool.

CONTACTS AND LOCATIONS:
Overall Officials: Earlise Ward, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No